CLINICAL TRIAL: NCT06575179
Title: Effect of Dexmedetomidine on Sevoflurane Minimum Alveolar Concentration for Attenuating Adrenergic Response to CO2 Pneumoperitoneum: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Reduces Sevoflurane MAC-BAR During Pneumoperitoneum
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: k2022-12-004
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: dexmedetomidine; MAC-BAR; sevoflurane; laparoscopic surgery; α2-adrenergic receptor agonist
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): The control group received volume-matched 0.9% saline infusions at identical rates.
  Interventions: Drug: normal Saline
- Low-dose dexmedetomidine group (Experimental): The low-dose dexmedetomidine group received a 75 μg/h loading dose over 15 minutes, followed by 60 μg/h maintenance infusion intravenously.
  Interventions: Drug: Dexmedetomidine low-dose
- High-dose dexmedetomidine group (Experimental): The high-dose dexmedetomidine group received a 150 μg/h loading dose over 15 minutes, followed by 120 μg/h maintenance infusion intravenously.
  Interventions: Drug: Dexmedetomidine high-dose

INTERVENTIONS:
Drug: Dexmedetomidine low-dose — The low-dose dexmedetomidine group received a 75 μg/h loading dose over 15 minutes, followed by 60 μg/h maintenance infusion intravenously.
  Other Names: dexmedetomidine hydrochloride Injection
  Arms: Low-dose dexmedetomidine group
Drug: normal Saline — The control group received volume-matched 0.9% saline infusions at identical rates.
  Arms: Control group
Drug: Dexmedetomidine high-dose — The high-dose dexmedetomidine group received a 150 μg/h loading dose over 15 minutes, followed by 120 μg/h maintenance infusion intravenously.
  Other Names: dexmedetomidine hydrochloride Injection
  Arms: High-dose dexmedetomidine group

SUMMARY:
This clinical trial aims to learn the impact of dexmedetomidine on the minimum alveolar concentration blunting the adrenergic response (MAC-BAR) of sevoflurane to carbon dioxide pneumoperitoneum in patients undergoing laparoscopic cholecystectomy. It will also learn about the effect of dexmedetomidine on hemodynamic parameters. The main questions are:

* Does dexmedetomidine reduce the MAC-BAR of sevoflurane required to suppress the sympathetic response to carbon dioxide pneumoperitoneum?
* Would dexmedetomidine administration dose-dependently reduce the minimum alveolar concentration blunting the adrenergic response of sevoflurane required to suppress the sympathetic response to carbon dioxide pneumoperitoneum? Researchers will compare low-dose dexmedetomidine to high-dose dexmedetomidine to see if dexmedetomidine works to treat postoperative negative behavior change and emergence delirium.

Participants will:

* Take intravenous dexmedetomidine or 0.9% saline (a look-alike substance that contains no drug)
* Study drug infusions were initiated 15 minutes prior to anesthesia induction, allowing a minimum of 30 minutes to elapse before surgical incision to achieve steady-state plasma and brain concentrations.

DETAILED DESCRIPTION:
Laparoscopic (minimally invasive) surgery has several advantages over open surgery, including less tissue damage, faster recovery, and fewer complications. This has led to widespread use of laparoscopic techniques. However, the inflated carbon dioxide gas used to create the surgical space during laparoscopic surgery causes significant changes in the body's normal blood pressure and heart function.

The anesthetic drug sevoflurane is commonly used during these procedures, but higher doses are needed to adequately block the body's stress response to the inflated gas. The minimum alveolar concentration blunting the adrenergic response (MAC-BAR) measures the minimum anesthetic depth required to suppress the sympathetic/stress response in 50% of patients. Doctors use MAC-BAR values to help determine the appropriate anesthetic dose to maintain hemodynamic stability. Unfortunately, using higher sevoflurane doses to reach the necessary MAC-BAR increases the risk of low blood pressure, reduced heart function, and confusion after surgery.

The drug dexmedetomidine has properties that can help manage the body's stress response during surgery. Researchers wanted to see if dexmedetomidine could allow the use of lower, more stable doses of sevoflurane during laparoscopic procedures by reducing the body's reaction to the inflated gas.

The goal of this study was to evaluate how dexmedetomidine affects the MAC-BAR of sevoflurane needed to block the sympathetic/stress response to the inflated gas used in laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-45 years.
* 2. American Society of Anesthesiologists (ASA) grade I - II.
* 3. Patients undergoing elective laparoscopic cholecystectomy.

Exclusion Criteria:

* 1. Inability to provide informed consent;
* 2. History of chronic pain or substance abuse;
* 3. Pregnancy;
* 4. Body mass index (BMI) ≥ 30 kg/m2;
* 5. Known allergies to the study medications;
* 6. Intake of medications within the last 72 hours that potential interfere with the determination of the MAC-BAR;
* 7. Any other condition deemed exclusionary by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Minimum alveolar concentration of sevoflurane to block the adrenergic response (MAC-BAR) | Within 30 minutes after intubation
  The MAC-BAR of sevoflurane for each group was determined using an up-and-down sequential allocation technique. One minute after establishing a stable pneumoperitoneum, the sympathetic adrenergic response was evaluated by changes in heart rate and mean artery pressure from pre-insufflation baseline values. A positive response was defined as a ≥ 20% increase in either heart rate or mean artery pressure from baseline.

SECONDARY OUTCOMES:
Change in mean arterial pressure | Upon arrival in the operating room, at 3, 1 minutes before pneumoperitoneum and 1, 3 minutes after pneumoperitoneum
  Change in blood pressure was calculated as the difference between pre-pneumoperitoneum and post-pneumoperitoneum. Pre-pneumoperitoneum mean arterial pressure was averaged from 3 and 1 minutes baseline values, while post-pneumoperitoneum value was averaged over 1 and 3 minutes after establishing insufflation.
Change in heart rate | Upon arrival in the operating room, at 3, 1 minutes before pneumoperitoneum and 1, 3 minutes after pneumoperitoneum
  Change in blood pressure was calculated as the difference between pre-pneumoperitoneum and post-pneumoperitoneum. Pre-pneumoperitoneum heart rate was averaged from 3 and 1 minutes baseline values, while post-pneumoperitoneum value was averaged over 1 and 3 minutes after establishing insufflation.
Incidence of adverse events | Up to 24 hours postoperatively
  Adverse events such as bradycardia, tachycardia, hypertension, hypotension, and hypoxia will be recorded during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD&PhD, Study Chair — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the individual deidentified participant data underlying published results, the study protocol, and the statistical analysis plan can be accessed upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The investigators would like to share the individual deidentified participant data from the three months following the publication of the main results.
Access Criteria: All the individual participant data collected during the trial, the study protocol, the statistical analysis plan, and the clinical study report can be accessed with approval from the corresponding author.